CLINICAL TRIAL: NCT06828965
Title: Neutrophil-Creatinine Index in Patients with Acute Pancreatitis: Assessment of Severity and Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Mohamed Abdelrahman, Principal Investigator Marwa Ahmed Mohamed Abdelrahman, Assiut University
Other Study IDs: Marwa protocol
Record Dates: First submitted 2025-01-27; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Acute Pancreatitis (AP)
Keywords: acute pancreatitis, severity, accuracy, mortality
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Neutrophil creatinine index — Neutrophil creatinine index will be calculated
Other: Neutrophil creatinine index — Neutrophi creatinine index will be calculated in all patients

SUMMARY:
Acute pancreatitis is a disease that usually has a mild disease course. However, around 20-30% of the patients develop severe complications. Persistent organ failure, with or without the presence of local complications such as (peri-) pancreatic necrosis and secondary infections, is the main determinant for mortality, and these patients are classified as having severe acute pancreatitis according to the revised Atlanta classification . The most widely used classification systems for determining the severity and course of AP are the revised Atlanta classification and the Bedside Index of Severity in Acute Pancreatitis (BISAP). According to the revised Atlanta classification, the severity of AP is graded as mild acute pancreatitis (MAP), moderately severe acute pancreatitis (MSAP), or severe acute pancreatitis (SAP) . In addition to the revised Atlanta classification and BISAP, several other prognostic scoring systems and classifications have been developed to predict the severity of AP. Ranson's criteria, the Acute Physiology and Chronic Health Evaluation (APACHE) II score, the Modified Glasgow Prognostic Score, and the Balthazar index are other commonly used prognostic systems . Most of these scoring systems include multiple determinants or parameters that must be noted 24 to 48 h after hospitalization, and the estimation of the severity of AP is delayed until 48 h after hospitalization. Thus, these scoring systems are of limited use at admission. On the other hand, in view of the complexity of prognostic scoring systems, several studies have been conducted on the role of simple laboratory parameters and indices in predicting the disease severity of AP and mortality . The most widely studied laboratory parameters and indices are the white blood cell count (WBC), neutrophil count, neutrophil to lymphocyte ratio (NLR), platelet to lymphocyte ratio (PLR), C-reactive protein (CRP), and procalcitonin. These laboratory parameters have also been used as part of several prognostic scoring systems. Nevertheless, none of the laboratory parameters or prognostic scoring systems can predict the severity of AP or MOF with sufficient accuracy . Moreover, it is not easy to predict the course and severity of acute pancreatitis at the first assessment of hospital admission. At the time of admission, most laboratory parameters are insufficient to differentiate mild disease from severe disease, and changes in laboratory parameters over time, including inflammatory markers and parameters related to organ/system dysfunction, provide important clues regarding the course of the disease . On the other hand, there is a need for simple, reliable, widely used parameters at admission for predicting the course of the disease. Sahin (2024) found a new index named the neutrophil-creatinine index (NCI), which was established based on the levels of neutrophil count and creatinine, to predict the severity of AP at admission . It's known that neutrophil infiltration and activation is one of the early events in acute pancreatitis and results in higher neutrophil count values at admission. Similarly, higher creatinine values at admission indicate renal hypoperfusion, which is associated with third-space leakage resulting from a systemic inflammatory state. It was assumed that the NCI may serve as an efficient test to represent the combination of inflammatory response and organ dysfunction .

DETAILED DESCRIPTION:
Inclusion criteria

* All patients with AP will be enrolled.
* Both sexes
* Age of patient > 18 years old Exclusion criteria Any patient with one or more of the following criteria is excluded;
* Age less than 18 years old
* Pancreatic cancer
* Picture of chronic pancreatitis
* Recurrent pancreatitis

ELIGIBILITY:
Inclusion Criteria:

* All patients with AP will be enrolled.
* Both sexes
* Age of patient > 18 years old

Exclusion Criteria:

* Age less than 18 years old
* Pancreatic cancer
* Picture of chronic pancreatitis
* Recurrent pancreatitis
* pregnancy, end-stage renal disease, hematological disorders, pancreatic carcinoma or cholangiocarcinoma, and incomplete records.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Based on previous reported estimated proportion of severe acute pancreatitis that was 15-20% (Silva-Vaz et al., 2020, Heckler et al., 2021) in addition to probability error 5% and 80% power on a two-tailed test, a minimum of 84 patients with acute pancreatitis are needed as an effective sample size for the current issue. To avoid drop out, a total of 120 patients will be recruited. It was calculated by OpenEpi
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-27 (Estimated); Primary Completion 2025-12-27 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of neutrophil/creatinine index in prediction severity of acute pancreatitis | One year
  A receiver operator characteristics curve will be used to determine the cut-off point of neutrophil/creatinine index in prediction severity of acute pancreatitis

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Ahmed Abdelrahman, Master Degree, Principal Investigator — Marwa Ahmed Abdelrahman
Locations (1):
- Assiut University Egypt, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Till finishing the study